CLINICAL TRIAL: NCT05103007
Title: A Multicenter, Randomized, Positive Parallel Controlled Clinical Trial of PVE/PVL Combined With DEB-TACE in the Treatment of Large or Large Liver Cancer in the Right Lobe of the Liver Without Hepatectomy
Brief Title: PVE/PVL Combined With DEB-TACE in the Treatment of Patients With Large and Unresectable Liver Cancer
Acronym: CCGLC-004
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, Prof., Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20210118
Record Dates: First submitted 2021-10-28; First posted 2021-11-02 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Drug-eluting bead transarterial chemoembolization(DEB-TACE); portal vein embolization(PVE); portal vein ligation(PVL)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-eluting bead transarterial chemoembolization（DEB-TACE) (Active Comparator): Percutaneous drug-eluting bead transarterial chemoembolization, followed by conventional transarterial chemoembolization（cTACE) every 2 months. A total of 3 times of chemoembolization will be performed.
  Interventions: Procedure: DEB-TACE
- PVL/PVE+DEB-TACE (Experimental): PVL and PVE will be performed randomly assigned according to 1:1 according to the random number table.
  Interventions: Procedure: PVL/PVE+DEB-TACE

INTERVENTIONS:
Procedure: DEB-TACE — It is suggested that the tumor feeding artery should be selected for the microcatheter. The mixed volume of pirarubicin 80mg + microsphere 2g is about 2ml, and the mixture of at least 10ml and contrast medium is slowly injected with 5-10min.
  Arms: Drug-eluting bead transarterial chemoembolization（DEB-TACE)
Procedure: PVL/PVE+DEB-TACE — DEB-TACE will be performed after the liver function recovered within 7-10 days. After that, conventional transarterial chemoembolization（cTACE) was performed every 2 months, a total of 2-3 times of chemoembolization.
  Arms: PVL/PVE+DEB-TACE

SUMMARY:
This is a multicenter, randomized, positive parallel controlled clinical study to evaluate the short-term and long-term efficacy and safety of PVL/PVE combined with DEB-TACE in the treatment of unresectable patients with large or large tumors in the right lobe of the liver.

DETAILED DESCRIPTION:
Most guidelines recommend transarterial chemoembolization (TACE) as the standard of treatment for hepatocellular carcinoma（HCC）which is limited to the right half of the liver, single large or multiple, with / without tumor thrombus of the right branch of the portal vein.While a number of studies demonstrate poor effect of TACE for patients with large hepatocellular carcinoma. Portal vein embolization(PVE)/portal vein ligation(PVL) is the main means to increase the future liver remnant (FLR), which can reduce the complications after hepatectomy. TACE on the basis of PVE/PVL can not only increase FLR, but also can effectively control the progression of tumor by sequential TACE. This study intends to conduct a multicenter, randomized, positive parallel-controlled clinical study to objectively and scientifically evaluate the short-term and long-term efficacy and safety of ligation of the right portal vein combined with Drug-eluting bead transarterial chemoembolization(DEB-TACE) technique in the treatment of patients with large or large tumors of the right lobe who cannot be resected in I-stage.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as large or giant hepatocellular carcinoma of the right lobe of the liver;
* Child-Pugh liver function grade A,
* ECOG PS 0-1
* If the tumor is resected with R0, the remaining liver volume is insufficient
* ICG-15R < 30%
* No serious organic diseases of heart, lung, brain and other organs;
* No history of other malignant tumors;
* The patient's survival time is expected to be more than 3 months.

Exclusion Criteria:

* Pregnant and lactating women
* History of organ transplant
* Tumor thrombus with portal vein trunk or left branch involved;
* distant metastasis;
* Patients with obvious liver cirrhosis (Plt < 100 × 10 ^ 9 / L at admission or gastroscopy suggested esophageal and gastric varices);
* Active bleeding caused by various causes;
* Suffering from severe acute or chronic diseases or infectious diseases;
* History of hepatectomy or TACE treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
the rate of tumor resection after treatment | Until one month after the last treatment.
FLR | Until one month after the last treatment.
  the ratio of FLR proliferation after treatment

SECONDARY OUTCOMES:
Overall survival (OS) | After operation, up to 3 years
  The overall survival time refers to the time from the first interventional therapy to the patient's death or the last follow-up, whichever appears early.
Progression-free survival (PFS) | 1, 3 year
  Disease progression-free survival time refers to the imaging evaluation of the patient after the first interventional therapy, the tumor does not continue to grow, new, distant metastasis; there is no increase in alpha-fetoprotein

CONTACTS AND LOCATIONS:
Overall Officials: Wan-guang Zhang, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China